CLINICAL TRIAL: NCT02927327
Title: Clinical Evaluation Of MP26 Features in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 114.03-2016-GES-0001
Record Dates: First submitted 2016-10-04; First posted 2016-10-07 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Brain Imaging; Whole Body Imaging
MeSH Terms: interventions — Radionuclide Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PET/MR ZTE MRAC (Experimental): PET/MR zero echo time (ZTE) scan for head attenuation and Q.Static . PET/MR ZTE MRAC images to be acquired for post-processing and reader assessment.
  Zero Echo Time (ZTE) scan for head attenuation
  Interventions: Device: Zero Echo Time (ZTE) scan for head attenuation
- PET/MR Q Static (Q. MRAC) (Experimental): Q.Static (Q. MRAC) for respiratory motion correction. PET/MR Q Static (Q. MRAC) images to be acquired for post-processing and reader assessment.
  PET/MR Q Static (Q. MRAC)
  Interventions: Device: Q.Static (Q. MRAC) for respiratory motion correction

INTERVENTIONS:
Device: Zero Echo Time (ZTE) scan for head attenuation — The GE SIGNA PET/MR MP26 software platform includes the zero echo time (ZTE) scan for head attenuation and Q.Static. The ZTE MR software feature has the potential to enable better visualization of bones, including those in the head, by employing optimal head attenuation correction in PET/MR.
  PET/MR ZTE MRAC
  Arms: PET/MR ZTE MRAC
Device: Q.Static (Q. MRAC) for respiratory motion correction — An improved Q.Static feature with Q. MRAC, where phase matching the MRAC with the quiescent phase is employed to get more accurate attenuation correction for our Q.Static PET images.
  PET/MR Q Static (Q. MRAC)
  Arms: PET/MR Q Static (Q. MRAC)

SUMMARY:
The purpose of the study is to collect representative clinical images (head and whole-body scans) of demonstrated diagnostic quality using the next-generation SIGNA PET/MR device equipped with investigational software components in adult population. The images and summary data from this study are intended for use in regulatory submission.

DETAILED DESCRIPTION:
Primary Objective: To demonstrate diagnostic image quality of image sets with ZTE MRAC and Q Static (Q. MRAC) for SIGNA PET/MR in representative clinical cases of the general imaging population.

Secondary Objective(s): To verify diagnostic acceptability, ease of use, and functionality of ZTE MRAC and Q Static (Q. MRAC) for SIGNA PET/MR at clinical sites.

Safety Objective(s): To collect information about safety events and device issues.

ELIGIBILITY:
Inclusion Criteria:

1. Are adults (aged 18 or older);
2. Have preexisting clinical indication for PET/CT or PET/MR with radiotracer injection (for subjects that will undergo ZTE procedures, a preexisting clinical indication for PET/CT is required);
3. Are able to undergo PET/MR within the tracer validity time frame after radiotracer injection;
4. Can hear without assistive devices and have necessary mental capacity to follow study instructions;
5. Are willing and able to provide written informed consent;
6. Are considered eligible for MRI and PET exams, according to site institutional safety policies.

Exclusion Criteria:

1. Were previously enrolled in the study;
2. If female, are pregnant or of undetermined pregnancy status;
3. Cannot fit safely in the device (>55 cm axial diameter or >227 kgs body weight);
4. Have implants or attached medical devices that could be unsafe for MRI;
5. Have medical conditions or require urgent care that could make it unsafe to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Duliskovich, M.D., Study Director — GE Healthcare, Medical Monitor
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PET/MR ZTE MRAC: PET/MR zero echo time (ZTE) scan for head attenuation and Q.Static . PET/MR ZTE MRAC images to be acquired for post-processing and reader assessment.
  Zero Echo Time (ZTE) scan for head attenuation
  Zero Echo Time (ZTE) scan for head attenuation: The GE SIGNA PET/MR MP26 software platform includes the zero echo time (ZTE) scan for head attenuation and Q.Static. The ZTE MR software feature has the potential to enable better visualization of bones, including those in the head, by employing optimal head attenuation correction in PET/MR.
  PET/MR ZTE MRAC
- PET/MR Q Static (Q. MRAC): Q.Static (Q. MRAC) for respiratory motion correction. PET/MR Q Static (Q. MRAC) images to be acquired for post-processing and reader assessment.
  PET/MR Q Static (Q. MRAC)
  Q.Static (Q. MRAC) for respiratory motion correction: An improved Q.Static feature with Q. MRAC, where phase matching the MRAC with the quiescent phase is employed to get more accurate attenuation correction for our Q.Static PET images.
  PET/MR Q Static (Q. MRAC)
Period: Overall Study
Arm/Group | PET/MR ZTE MRAC | PET/MR Q Static (Q. MRAC)
Started | 30 | 31
Completed | 30 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PET/MR ZTE MRAC | PET/MR Q Static (Q. MRAC) | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 11 | 28
  >=65 years | 13 | 20 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (12.86) | 67.3 (10.76) | 64.0 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 18 | 17 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Image Quality
Description: scored on a 5-pt Likert scale:
  1. Unacceptable
  2. Poor
  3. Acceptable
  4. Good
  5. Excellent
Time Frame: through study completion, an average of 2 months
Population: Subjects that had a clinical indication for PET/CT or PET/MR with radiotracer injection prescribed for their medical care outside of the study.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PET/MR ZTE MRAC | PET/MR Q Static (Q. MRAC)
Number analyzed (Participants) | 30 | 31
scores on a scale | 4.4 (0.54) | 3.9 (0.68)

2. Secondary Outcome: Determination of Diagnostic Acceptability
Description: Site level determination of diagnostic acceptability (Y/N) based on consensus between radiologist(s) and nuclear medicine physician(s) at the site. Diagnostic acceptability in the form of binary responses (Y/N) were collected from 61 subjects who completed the study.
Time Frame: through study completion, an average of 2 months
Population: Diagnostic acceptability in the form of binary responses (Y/N) were collected from 61 subjects who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | PET/MR ZTE MRAC | PET/MR Q Static (Q. MRAC)
Number analyzed (Participants) | 30 | 31
Participants | 30 | 31

3. Secondary Outcome: Ease of Use Per Procedure Rated on a 5-pt Likert Scale Score
Description: Ease of use ratings, based on a 5-point Likert scale (e.g. 1=unacceptable, 2=poor, 3=acceptable, 4=good, 5=excellent), were collected from the population of subjects who completed the study.
Time Frame: through study completion, an average of 2 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | PET/MR ZTE MRAC | PET/MR Q Static (Q. MRAC)
Number analyzed (Participants) | 30 | 31
scores on a scale
  Prescribing PET scan | 4.6 (0.73) | 4.6 (0.73)
  Prescribing MR scans simultaneous with PET | 4.6 (0.73) | 4.6 (0.73)
  Starting and monitoring scanning | 4.6 (0.81) | 4.6 (0.81)
  Reviewing PET and MR images | 4.6 (0.73) | 4.6 (0.73)
  Overall process of doing this exam | 4.6 (0.78) | 4.6 (0.78)
  Performing exam within acceptable duration to meet | 4.6 (0.85) | 4.6 (0.85)

4. Secondary Outcome: Number of Participants Reporting "Yes" On All Binary Performance Scale Questions
Description: The number of participants reporting "yes" on a binary performance scale (Y/N) were collected.
Time Frame: through study completion, an average of 2 months
Population: Functionality ratings, based on a binary performance scale (Y/N), were collected from the population of subjects who completed the study, including both ZTE and Q.Static populations (N=61 total subjects).
Measure: Count of Participants; unit: Participants
Arm/Group | PET/MR ZTE MRAC | PET/MR Q Static (Q. MRAC)
Number analyzed (Participants) | 30 | 31
Participants | 30 | 31

5. Other Pre Specified Outcome: Summary of Safety Information
Description: Number of safety events (AEs and SAEs).
Time Frame: through study completion, an average of 2 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from the time the subject entered the PET/MR suite until the subject left the PET/MR suite, an average of less than 2 hours.
Arm/Group | PET/MR ZTE MRAC | PET/MR Q Static (Q. MRAC)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT02927327/Prot_SAP_000.pdf